CLINICAL TRIAL: NCT06180213
Title: Study of Cerebral Glucose Metabolism in Neurodegenerative Diseases and Head Trauma: Retrospective Review of an Large Cohort of FDG PET Data
Brief Title: Study of Cerebral Glucose Metabolism in Neurodegenerative Diseases and Head Trauma
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: FDG-PET
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FDG PET — Distribution pattern of the FDG tracer in patients with neurodegenerative diseases and identify the regions of altered brain function specific for each clinical condition.

SUMMARY:
The reason why each specific degenerative disease is characterized by a different FDG PET pattern is still unclear today. There are four main hypotheses proposed to explain this selective vulnerability: 1) Nodal stress, theory according to which the main nodes of specific brain networks undergo wear and tear, 2) trans-neuronal diffusion, theory according to which some toxic agents/proteins or altered propagate along network connections through "Prion-like" mechanisms, 3) trophic failure, in which the interruption of inter-modal connectivity causes the loss of collateral trophic factors, and finally 4) shared vulnerability in which regions also distant from each other are part of a common network which gives a susceptibility uniformly distributed throughout the network.

FDG PET provides in-vivo information on the distribution of brain synaptic dysfunction prior to complete neural death, and represents the main in vivo biomarker of neural dysfunction associated with different clinical conditions characterized by neurodegeneration phenomena. For this reason, FDG PET is considered a fundamental approach to shed light on the causes of selective brain vulnerability in various pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

* presence of diagnosis of neurodegenerative disease.

Exclusion Criteria:

* patients< 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients suffering from various forms of Alzheimer's dementia, Parkinsonism, ALS, motor neuron diseases.
Sampling Method: Probability Sample
Enrollment: 1570 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
FDG PET to measure brain areas of hypo or hyper regional metabolism in patients with neurodegenerative disease. | 4 years
  Characterization of the different pathologies examined starting from the study of regional metabolism in individual subjects up to the study of the functional activity of the different brain circuits.

IPD SHARING:
Plan to Share IPD: No